Evrak Tarih ve Sayısı: 19.10.2022-E.487579



## GAZİ ÜNİVERSİTESİ REKTÖRLÜĞÜ **Etik Komisyonu**

E-77082166-604.01.02-487579 19.10.2022 Sayı:

Konu: Değerlendirme ve Onay

## Sayın Doç.Dr. Zait Burak AKTUĞ Niğde Ömer Halisdemir Üniversitesi Spor Bilimleri Fakültesi

Araştırmacı grubu Zait Burak AKTUĞ, Serkan İBİŞ, Cengiz AKARÇEŞME, Hasan AKA, Bökebatur Ahmet Raşit MENDİ, Necdet Eray PİŞKİN, Gönül YAVUZ ve oluşan "Kan Akışı Kısıtlama Yöntemi ile Kombinlenen Düşük Yoğunluklu Bisiklet Egzersizlerinin MaxVO2, Kas Kuvveti ve Kas Kalınlığına Etkisi'' başlıklı araştırma öneriniz Komisyonumuzun **04.10.2022** tarih ve **16** sayılı toplantısında görüşülmüş olup,

Çalışmanızın, yapılması planlanan yerlerden izin alınması koşuluyla yapılmasında etik açıdan bir sakınca bulunmadığına oybirliği ile karar verilmiş ve karara ilişkin imza listesi ekte gönderilmiştir.

Bilgilerinizi rica ederim.

Araştırma Kod No: 2022 - 961

Prof. Dr. Fazlı POLAT Rektör Yardımcısı

Ek:1 Liste

Bu belge, güvenli elektronik imza ile imzalanmıştır.

Belge Takip Adresi: https://www.turkiye.gov.tr/gazi-universitesi-ebys







Evrak Taril<del>ı ve Sayısı: 19.10.2022-E.487579</del> GAZİ ÜNİVERSİTESİ
ETİK KOMİSYONU KATILIM LİSTESİ

| TOPLANTI TARİHİ : 04.10.2022 | TOPLANTI SAYISI : 16 | |
|-------------------------------------|----------------------|---|
| ADI – SOYADI | | |
| Prof. Dr. İsmail KARAKAYA<br>BAŞKAN | | |
| Prof.Dr.C.Haluk BODUR | | |
| Prof.Dr.Seçil ÖZKAN | 5 | |
| Prof.Dr.Cevriye TEMEL GENCER | К | |
| Prof.Dr.İsmet YÜKSEL | ( | |
| Prof.Dr.Aymelek GÖNENÇ | | |
| Prof.Dr.Gülay BAYRAMOĞLU | | |
| Prof.Dr.Makbule GEZMEN KARADAĞ | N | ( |
| Prof.Dr.Zehra GÖÇMEN BAYKARA | | |
| Prof.Dr.İlyas OKUR | | _ |
| Prof.Dr.Nihan KAFA | | |
| Doç.Dr.Melek Gülşah ŞAHİN | | |